CLINICAL TRIAL: NCT00452829
Title: Prevention of Neural Tube Defects by Inositol in Conjunction With Folic Acid (PONTI Study)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institute of Child Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 05ND07
Record Dates: First submitted 2007-03-27; First posted 2007-03-28 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Recurrent Neural Tube Defects
MeSH Terms: conditions — Neural Tube Defects | interventions — Folic Acid; Inositol; Control Groups

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study Group (Experimental): 5 mg folic acid (the standard UK supplement for pregnancies at high risk of NTD) and 1 g inositol,
  Interventions: Drug: Folic Acid and inositol
- Control Group (Placebo Comparator): 5 mg folic acid (the standard UK supplement for pregnancies at high risk of NTD)and 1 g placebo
  Interventions: Drug: Folic acid and placebo

INTERVENTIONS:
Drug: Folic Acid and inositol — Folic Acid and inositol
  Other Names: Study Group
  Arms: Study Group
Drug: Folic acid and placebo — Folic acid and placebo
  Other Names: Control Group
  Arms: Control Group

SUMMARY:
The aim of the study is to develop a randomised, double blind clinical trial to compare (i) folic acid plus inositol, with (ii) folic acid plus placebo, for prevention of recurrent neural tube defects.

DETAILED DESCRIPTION:
Women were eligible to join the PONTI pilot study if they had a history of previous NTD-affected pregnancy, were planning to become pregnant again, and were prepared to be randomised to one of the two study arms. Both study and control groups received 5 mg folic acid (the standard UK supplement for pregnancies at high risk of NTD); the study group additionally received 1 g inositol, whereas the control group was prescribed a placebo instead of inositol.

ELIGIBILITY:
Inclusion Criteria

1. Women with a history of one or more NTD pregnancies (spina bifida, anencephaly or encephalocele) who wished to embark upon a further pregnancy.

Exclusion criteria

1. Women who were unable to give informed consent for any reason (language difficulties, low IQ).

   Funding was not available to translate the information leaflets or to employ interpreters for the telephone interviews. It was intended to take appropriate measures to include these groups in a definitive follow-up trial.
2. Maternal age outside 18 - 40 years of age. An upper limit of forty years was stipulated because there is increased risk of a pregnancy being affected by chromosomal abnormality which may result in a NTD, but which may not be similarly susceptible to prevention by nutrient supplementation.
3. Cases where the previous affected child had abnormalities other than NTD, which might be suggestive of another underlying genetic aetiology, a chromosomal abnormality or fetal valproate syndrome. In these cases the underlying pathology would be different from spontaneous, isolated NTDs, and folic acid or inositol would not be expected to influence recurrence risk.
4. Women who were epileptic and/or taking anti-epileptic medications including valproate. It was recognised that some anti-epileptic drugs increase the predisposition to NTDs and, such NTDs might be unresponsive to inositol supplementation.
5. Women who did not have a GP or obstetrician in the UK. We needed to be able to monitor the pregnancy, confirm there were no contraindications to inositol supplementation, and seek outcome data. We did not have the facilities to seek this information for cases outside the UK.
6. Women would be required to stop participation in the trial if the following criteria were met whilst taking the prescribed drugs;

   * Diagnosed with epilepsy and were therefore required to take anti-epileptics.
   * Failed to conceive within one year of starting the trial.
   * They no longer wished to conceive .

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2009-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Copp, Prof, Principal Investigator — Institute Of Child Health and Great Ormond Street Hospital
Locations (1):
- Neural Development Unit, Institute of Child Health, London, United Kingdom